CLINICAL TRIAL: NCT02326961
Title: Celution Prepared Adipose Derived Regenerative Cells in the Treatment of Osteoarthritis of the Knee: A Double-blind, Placebo Controlled, Multi-center Safety and Feasibility Study
Brief Title: Celution Prepared Adipose Derived Regenerative Cells in the Treatment of Osteoarthritis of the Knee
Acronym: ACT-OA Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT-OA Knee
Record Dates: First submitted 2014-11-19; First posted 2014-12-30 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; adipose derived regenerative cells; ADRC; Celution; arthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Celution ADRCs; Low Dose (Experimental): Adipose Derived Regenerative Cells (ADRCs) processed by the Celution Device 20,000,000 ADRCs per single intraarticular administration
  Interventions: Device: Celution Device
- Celution ADRCs; High Dose (Experimental): Adipose Derived Regenerative Cells (ADRCs) processed by the Celution Device 40,000,000 ADRCs per single intraarticular administration
  Interventions: Device: Celution Device
- Placebo (Placebo Comparator): Sterile Lactated Ringers Solution (5mL) mixed with ≤ 0.20 ml of the study subject's own freshly drawn blood.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Celution Device — ADRCs Prepared using the Celution Device
  Arms: Celution ADRCs; High Dose; Celution ADRCs; Low Dose
Other: Placebo — Inactive Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and feasibility of intraarticular injection of Celution prepared adipose-derived regenerative cells injected into knees of patients with chronic knee pain due to osteoarthritis.

DETAILED DESCRIPTION:
The ACT - OA Knee Clinical Trial is a prospective, randomized, multi-center device trial intended to assess safety and feasibility of intraarticular administration of Celution processed Adipose Derived Regenerative Cells (ADRCs). The study will include 90 patients in up to 15 sites in the United States.

Subjects that have chronic knee pain due to idiopathic osteoarthritis of the knee (confirmed clinically and radiologically) will be evaluated for eligibility in this study. Following informed consent and screening evaluations, eligible subjects will undergo pre-operative testing. Subjects will then undergo fat harvest through small volume liposuction under local anesthesia. Lipoaspirate will be processed in the Celution System to isolate and concentrate ADRCs for immediate intraarticular administration. A dose escalation approach has been designed wherein the study is divided into two double-blind, randomized, placebo-controlled parts as follows:

Part A:

Low Dose (20,000,000 cells): 30 patients OR Placebo: 15 patients

Part B:

High Dose (40,000,000 cells): 30 patients OR Placebo: 15 patients

Subjects randomized to placebo will undergo fat harvest and intraarticular injection of a placebo that has been visually matched to the active test substance. All subjects will undergo imaging studies, clinical evaluations, and laboratory testing prior to and after the procedure; patients will be followed for 48 weeks after intraarticular injections are performed.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 40 and < 70 years of age
2. Able to provide written informed consent
3. Diagnosis of osteoarthritis in one or both knees by American College of Rheumatology (ACR) criteria
4. Kellgren and Lawrence grade 2 or 3 (standing AP x-ray) of the target knee within the preceding 6 months
5. Pain due to osteoarthritis in the target knee ≥ 6 months
6. Minimum score of "moderate" from KOOS question about pain on walking on a flat surface.
7. Minimum score of "moderate" from KOOS question about degree of difficulty during walking on a flat surface.
8. Continued knee pain and limitations in knee function despite prescription of conservative therapy for at least 6 months.
9. Ability to safely undergo liposuction that will result in the harvest of a sufficient quantity of adipose tissue (approximately 300 mL)
10. On stable regimen of one analgesic medication (rescue medication) for their knee pain due to osteoarthritis and ability and willingness to use the same analgesic medication during the study (screening period through to final study visit).
11. Ability to perform procedures required of the pain index evaluations (unassisted walking 50 feet on a flat surface and going up and down stairs)

Exclusion Criteria:

1. Any major injury to the target knee within the 12 months prior to the screening visit
2. Need for cane or other assistance device for walking
3. Any surgery to the target knee within the 6 months prior to the screening visit, or surgery to the contralateral knee or other weight-bearing joint if it will interfere with knee assessments
4. Prior articular transplant procedures
5. Prior ligament reconstruction to the target knee within 12 months prior to the screening visit
6. Inflammatory arthropathies such as rheumatoid arthritis, lupus arthropathy, or psoriatic arthritis
7. Gout or calcium pyrophosphate (pseudogout) diseases that have flared within the previous 6 months prior to the screening visit
8. X-ray findings of acute fractures, known severe loss of bone density (as determined by the investigator), avascular necrosis, and/or severe bone or joint deformity in the target knee (>5 degree valgus or varus deviation from mechanical axis)
9. Fibromyalgia, pes anserine bursitis, lumbar radiculopathy, and/or neurogenic or vascular claudication
10. Primary knee pain due to diagnosed isolated patella-femoral arthritis or chondromalacia in the target knee
11. Significant target knee joint infection or skin disorder/infection within the previous 6 months prior to the screening visit
12. Symptomatic OA of the hips, spine, or ankle, if it would interfere with the evaluation of the target knee
13. Any condition requiring immunosuppressive medication or use of systemic steroids
14. Intra-articular injection of steroids in previous 3 months or hyaluronic acid in previous 6 months in one or both knees prior to the screening visit
15. Patients that have received PRP, other platelet-based product, or investigational treatment in another cell/biologic study for the targeted treatment injury in the 12 months prior to the injection procedure
16. Participation in any experimental drug or device study within the 6 months prior to the screening visit
17. Obesity defined as BMI > 35 kg/m2

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) - Pain on Walking | 12 Weeks

SECONDARY OUTCOMES:
Observed Pain Scores on 50-foot Walk Test | 48 Weeks
Number of Observed OARS130 Responders | 48 Weeks
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 48 Weeks
VAS Assessments | 48 Weeks
Patient Global Assessment | 48 Weeks
Use of Rescue Medication | 48 Weeks
SF-36 Questionnaire | 48 Weeks
MRI Osteoarthritis Knee Score | 48 Weeks

OTHER OUTCOMES:
Adverse Events, Serious Adverse Events, and UADEs | 48 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, MD, Study Director — Cytori Therapeutics
Locations (11):
- United States (11):
  - Arizona Arthritis and Rheumatology Research, PLLC, Mesa, Arizona
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - BioSolutions Clinical Research Center, La Mesa, California
  - Rush University Medical Center, Chicago, Illinois
  - Heartland Research Associates, Wichita, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Covington Orthopedic and Sports Medicine Institute, Covington, Louisiana
  - Arthritis Treatment Center, Frederick, Maryland
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Hospital for Special Surgery, New York, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania